CLINICAL TRIAL: NCT07010809
Title: Assessing Bone Thermal Damage in Knee Arthroplasty: Burring vs Sawing
Brief Title: Comparing Temperature in Burr vs Saw Cutting for Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23/015
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic Total Knee Arthroplasty: With burr cutting
- Conventional Total Knee Arthroplasty: With saw cutting

SUMMARY:
We will assess the temperatures achieved during bone cutting in total knee replacements, comparing burr and saw techniques. Our study involves recruiting 20 patients from East Suffolk and North Essex NHS Foundation Trust (Colchester site). Patients will be recruited from the orthopaedic outpatient clinic, with 10 undergoing Robotic total knee arthroplasty (burr cutting) and 10 undergoing conventional total knee arthroplasty (saw cutting). Temperatures will be measured using a visual infrared thermometer placed outside the surgical field while a consultant surgeon performs the procedure. Importantly, these temperature recordings will have no impact on which treatment the patient received as the standard of care.

DETAILED DESCRIPTION:
Patients will be recruited from elective orthopaedic outpatient clinics. All patients over the age of 18 with symptomatic osteoarthritis (OA), and due to undergo robotic assisted rTKA, with burr cutting, or cTKA, with saw cutting, will be considered for trial inclusion. Both devices are considered the standard of care for TKA.

This is an observational trial and the decision to undergo rTKA or cTKA is determined by patient factors, availability of equipment, and following consultation with the surgeon. The trial will not influence which patients undergo rTKA or cTKA.

10 patients undergoing cTKA and 10 patients undergoing rTKA will be recruited. During the procedure, a thermal imaging camera (Thermovision A320, Flir Systems Inc., Wilsonville, Oregon, USA) will be setup 2 metres outside the sterile operating field to record temperatures reached during the distal femoral cut.

* Patients diagnosed with osteoarthritis follow a streamlined pathway to consult an orthopaedic surgeon. Initially, during the first clinic visit, the diagnosis is verified through both imaging and clinical examinations. After confirming the diagnosis, the patient is then scheduled for surgery, which could be either a robotic-assisted or a conventional total knee replacement, depending on their needs.
* Approximately 1-2 weeks prior to the surgery, patients attend a consent clinic. During this session, if they meet the inclusion criteria, they are provided with detailed study information and invited to participate. For those needing more time to decide, the option to take the consent form home is available. This gives them at least 1-2 weeks to consider their enrolment before the surgery.
* This study will not in any way impact the high standard of care provided to our patients. It is essential for researchers to ensure that enrolled patients have a comprehensive understanding of the trial procedures, the utilization of pseudo anonymized data, and contact addresses for any questions.
* The study includes no direct intervention- it is an observational study.
* A thermal imaging camera (Thermovision A320, Flir Systems Inc., Wilsonville, Oregon, USA) will be used to monitor temperature at the bone interface from exposure of distal femur until the distal femoral cut has been completed.
* The camera will be positioned 2 meters away from the operative site out of the sterile operating field and will be operated by a trained members of staff who are members of the direct clinical care team.
* All measurements throughout the study will be captured with the same camera, calibrated to the ambient room temperature and humidity prior to use in accordance with the manufacturer's instructions.
* The camera will be connected to a password protected ESNEFT laptop computer, running the software application required to control and record from the thermal imaging camera (ThermaCAM Researcher Pro, version 2.8, Flir Systems Inc., Wilsonville, Oregon, USA, http://www.flir.com/).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis
* 18+ years old
* Scheduled for TKA as part of standard of care

Exclusion Criteria:

* Distorted bone anatomy
* Previous knee surgery
* Diagnosed disease affected bone quality (e.g. Rheumatoid arthritis, Paget's disease, Osteomalacia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to Colchester hospital for a total knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The measure of temperature generated by burr and saw cutting devices during total knee arthroplasty. | During surgery
  Temperature will be measured in degrees centigrade

SECONDARY OUTCOMES:
Duration of temperature above 47 degrees centigrade in burr and saw cutting groups. | During surgery.
  Temperature will be measured in degrees centigrade.

CONTACTS AND LOCATIONS:
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Colchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Results of the temperatures recorded by the device will be published in peer-reviewed scientific journals and conference presentations.